CLINICAL TRIAL: NCT05625620
Title: A Long Term At-home Trial With Cerebellar-spinal Transcranial Pulsed Current Stimulation (tPCS) for Treatment of Neurodegenerative Ataxia
Brief Title: Cerebellar-spinal Transcranial Pulsed Current Stimulation (tPCS) for Treatment of Neurodegenerative Ataxia
Acronym: tPCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Mandar Jog, Professor, Western University, Canada
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 121665
Record Dates: First submitted 2022-11-01; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Cerebellar Ataxia
Keywords: Non-invasive Stimulation; Transcranial Pulsed Current stimulation
MeSH Terms: conditions — Cerebellar Ataxia

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Real tPCS (Experimental): All patients will be randomized into daily cerebello- spinal tPCS or sham stimulation. Randomization will occur in a ratio of 1:1. Real tPCS arm will receive active tPCS. Then they will be crossed over to Sham tPCS arm.
  Interventions: Device: Active Transcranial Pulse Current Stimulation
- Sham tPCS (Experimental): All patients will be randomized into daily cerebello- spinal tPCS or sham stimulation. Randomization will occur in a ratio of 1:1. Sham tPCS arm will receive active tPCS. Then they will be crossed over to Real tPCS arm.
  Interventions: Device: Sham Transcranial Pulse Current Stimulation

INTERVENTIONS:
Device: Active Transcranial Pulse Current Stimulation — Active tPCS will be delivered through a pair of saline-soaked (0.9% NaCl) surface sponge electrodes (7 × 5 cm2, for the anodal cerebellar electrode; 8 × 6 cm2 for the cathodal spinal electrode). Anodal stimulation will be applied on the scalp over the cerebellum area (2 cm under the inion) and the cathode will be placed over the spinal lumbar enlargement (2 cm under T11). During anodal stimulation, a constant current of 2 mA will be applied for 20 minutes.
  Arms: Experimental: Real tPCS
Device: Sham Transcranial Pulse Current Stimulation — Sham tPCS will be delivered through a pair of saline-soaked (0.9% NaCl) surface sponge electrodes (7 × 5 cm2, for the anodal cerebellar electrode; 8 × 6 cm2 for the cathodal spinal electrode). Anodal stimulation will be applied on the scalp over the cerebellum area (2 cm under the inion) and the cathode will be placed over the spinal lumbar enlargement (2 cm under T11). During anodal stimulation, a constant current of 2 mA will be applied for 20 minutes. Electric Current will be ramped down 5 seconds after the beginning of the stimulation to make this condition indistinguishable from the experimental active stimulation.
  Arms: Sham tPCS

SUMMARY:
Neurodegenerative ataxia represents a group of disabling diseases. Patients mainly present with imbalance during walking, speech problem and difficulty in co-ordination during working with hands. No effective treatment is currently available for them. Currently, studies are going on the effectiveness of noninvasive brain stimulation (NIBS) in neurodegenerative diseases. It is a mode of brain stimulation technique where current is delivered into the brain by placing electrodes into their scalp. Transcranial pulsed current stimulation (tPCS) is a new modality of NIBS. . The clinical benefit observed after a single session of tPCS in 15 patients with neurodegenerative ataxia, suggest that prolonged stimulation could be even more effective. The investigator have planned to study the efficacy of long-term tPCS in these patients of neurodegenerative ataxia.

Patients will be first examined clinically by the researcher along with the Scale for the Assessment and Rating of Ataxia (SARA) and Cerebellar Cognitive Affective Syndrome Scale (CCAS). Upper limb motor function, speech and Gait will be assessed according to the established protocol.

After the screening visit and inclusion, all patients will be randomized into daily cerebello- spinal tPCS or sham stimulation.

Anodal stimulation will be used for cerebellum and cathodal stimulation for the spinal stimulation. 20 min of non-invasive stimulation will be given via tPCS either real or sham stimulation. Patients will be trained and tolerability and ability to self-administer tPCS at home will be determined. Patients will continue tPCS at home 20 min daily for 2 weeks (7 days/week for 2 weeks). Assessments will be carried out 2 weeks after the first intervention (either real or sham tPCS).Then, patients will be reassessed at 1-month and 3-months follow-ups. After a washout period of 3 months since the last visit, each patient will receive the opposite treatment and undergo the same standardized assessment as in the first phase.

DETAILED DESCRIPTION:
The investigator have planned to study the efficacy of long-term tPCS in these patients of neurodegenerative ataxia. Anodal stimulation will be used for cerebellum and cathodal stimulation for the spinal stimulation.

After the screening visit and inclusion, all patients will be randomized into daily cerebello- spinal tPCS or sham stimulation. Randomization will occur in a ratio of 1:1. After a washout period of three months, all patients will be crossover to the other intervention. By the end of the study all patients will receive a cycle of tPCS and a cycle of sham stimulation. Clinical rater will be blinded throughout the whole study.

After screening and randomization, all patients will undergo a baseline clinical assessment. A blinded researcher will apply the Scale for the Assessment and Rating of Ataxia (SARA) and the Cerebellar Cognitive Affective Syndrome Scale (CCAS). Also will asses speech, gait, and upper limb motor function. Speech will be assessed according to the established protocol. Gait will be assessed via Gait Carpet. Upper limb motor function will be assessed by a robotic arm called KinArm. At the initial visit, the patient will be trained and tolerability and ability to self-administer tPCS at home will be determined.Assessments will be carried out 2 weeks after the first intervention (either real or sham tPCS) .Then, patients will be reassessed at 1-month and 3-months follow-ups. After a washout period of 3 months since the last visit, each patient will receive the opposite treatment and undergo the same standardized assessment as in the first phase.

tPCS will be delivered through a pair of saline-soaked (0.9% NaCl) surface sponge electrodes (7 × 5 cm2, for the anodal cerebellar electrode; 8 × 6 cm2 for the cathodal spinal electrode). Anodal stimulation will be applied on the scalp over the cerebellum area (2 cm under the inion) and the cathode will be placed over the spinal lumbar enlargement (2 cm under T11). During anodal stimulation, a constant current of 2 mA will be applied for 20 minutes. For the sham condition, electrode position will be same, but the electric current will be ramped down 5 seconds after the beginning of the stimulation to make this condition indistinguishable from the experimental active stimulation.

Participant's speech will be recorded using a head-mounted microphone (AKG-c520) and a digital recording device (Zoom H4nPro) while performing the following calibrated tasks. Calibration involves a sound level meter placed at 15cm from the mouth while talker says 'ah' at 70dBA. The following speech tasks will be assessed-

1. Prolonged 'ah'.
2. Rapid repetitions of the sounds "puh", "tuh", and "kuh".
3. Two productions of a sentence with selected speech sounds (s, sh, p, b, t, i, a, u, ae, ai). "She saw Patty buy two poppies."
4. Two times louder production of a sentence with selected speech sounds. "She saw Patty buy two poppies."
5. Repetition of a continuous vowel at normal and fast rates. 'eye-eye-eye-eye-eye' without making any voice breaks or pauses".
6. Read aloud a section of a standard passage - standard rainbow passage
7. Monologue. Talk for two minutes about an interesting vacation (or an interesting hobby or activity).

For gait, the Zeno walkway it will be used. The Zeno walkway will be used in conjunction with the ProtoKinetics Movement Analysis Software (PKMAS). This detects pressure data during gait, balance, and additional movement protocols.

For measuring upper limb movements, KinARM will be used which is the short form of a robotic device. The KinARM initially provides the patients with multiple points to reach in the screen and the patients would try to reach these points using the KinARM handle.

All quantitative data will be expressed in term of medians and interquartile range. For qualitative variables, data will be expressed in total numbers and proportions (percentages).

Quantitative results from every assessment (T0, T1, T2 and T3) will be compared between sham and real stimulation using the Wilcoxon signed-rank test for paired samples. For qualitative data, variables will be compared using the chi-square (χ 2) test or the Fisher's exact test when appropriate. For all analyses a p<0.05 was specified as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with neurodegenerative ataxia (clinically or by genetic study).

Exclusion Criteria:

* Patients unable to walk even with support (wheelchair or bed bound patients for example)
* Other comorbidities deemed by the investigators to interfere with clinical, motor, gait or qEEG assessments.
* Patients with Pacemaker
* Patients with metal implants in the head/neck region
* Severe comorbidity
* Intake of illegal drugs
* Pregnancy
* Patients unable to provide informed consent
* Patients unable to communicate in English.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Scale for the Assessment and Rating of Ataxia (SARA) Score From Baseline after 2-week/daily tPCS | Baseline - 2 weeks - 1 month - 3 months
  The investigators will evaluate the effectiveness of tPCS in patients of neurodegenerative ataxia applying the Scale for the Assessment and Rating of Ataxia (SARA) pre and post stimulation. The scale is for assessing severity of ataxia, that consists of assessment of gait, stance, sitting, speech, finger chase, finger to nose test, fast alternating hand movement, heel-shin test. The total score ranges from 0( no ataxia) to 36(most severe ataxia).

SECONDARY OUTCOMES:
Changes in spatiotemporal gait measures using objective gait analysis | Baseline - 2 weeks - 1 month - 3 months
  The investigators will use Zeno Walkway Gait carpet and the spatiotemporal details of the gait will be analyzed by ProtoKinetics Movement Analysis Software (PKMAS) software, pre and post stimulation
Change in speech | Baseline - 2 weeks - 1 month - 3 months
  The investigators will use standardized speech protocol pre and post stimulation to assess speech
Change in upper limb co-ordination | Baseline - 2 weeks - 1 month - 3 months
  The investigators will use KinArm pre and post stimulation to have objective measurement of upper limb co-ordination
Change in the Cerebellar cognitive affective syndrome (CCAS) Scale From Baseline | Baseline - 2 weeks - 1 month - 3 months
  CCAS/Schmahmann syndrome scale: 120 point scale, yielding a total score of 0 (most severe cognitive impairment) to 120 (no cognitive impairment).

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Result] Manto M, Gandini J, Feil K, Strupp M. Cerebellar ataxias: an update. Curr Opin Neurol. 2020 Feb;33(1):150-160. doi: 10.1097/WCO.0000000000000774. PMID 31789706
- [Result] Kim JS, Cho JW. Hereditary Cerebellar Ataxias: A Korean Perspective. J Mov Disord. 2015 May;8(2):67-75. doi: 10.14802/jmd.15006. Epub 2015 May 31. PMID 26090078
- [Result] Benussi A, Pascual-Leone A, Borroni B. Non-Invasive Cerebellar Stimulation in Neurodegenerative Ataxia: A Literature Review. Int J Mol Sci. 2020 Mar 12;21(6):1948. doi: 10.3390/ijms21061948. PMID 32178459
- [Result] Benussi A, Dell'Era V, Cotelli MS, Turla M, Casali C, Padovani A, Borroni B. Long term clinical and neurophysiological effects of cerebellar transcranial direct current stimulation in patients with neurodegenerative ataxia. Brain Stimul. 2017 Mar-Apr;10(2):242-250. doi: 10.1016/j.brs.2016.11.001. Epub 2016 Nov 3. PMID 27838276
- [Result] Ganguly J, Murgai A, Sharma S, Aur D, Jog M. Non-invasive Transcranial Electrical Stimulation in Movement Disorders. Front Neurosci. 2020 Jun 5;14:522. doi: 10.3389/fnins.2020.00522. eCollection 2020. PMID 32581682
- [Result] Alon G, Yungher DA, Shulman LM, Rogers MW. Safety and immediate effect of noninvasive transcranial pulsed current stimulation on gait and balance in Parkinson disease. Neurorehabil Neural Repair. 2012 Nov-Dec;26(9):1089-95. doi: 10.1177/1545968312448233. Epub 2012 May 10. PMID 22581566
- [Result] Benussi A, Dell'Era V, Cantoni V, Bonetta E, Grasso R, Manenti R, Cotelli M, Padovani A, Borroni B. Cerebello-spinal tDCS in ataxia: A randomized, double-blind, sham-controlled, crossover trial. Neurology. 2018 Sep 18;91(12):e1090-e1101. doi: 10.1212/WNL.0000000000006210. Epub 2018 Aug 22. PMID 30135258